CLINICAL TRIAL: NCT06836674
Title: The Effects of Three Different Methods (Metaverse, Jigsaw, Classical) on Students' Self-efficacy Levels in Pediatric Drug Administration
Brief Title: Pediatric Drug Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Şerife TUTAR GÜVEN, Assisstant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 72867572-050.01.04-87
Record Dates: First submitted 2024-08-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Nursing; Drugs, Investigational
Keywords: Pediatric Nursing; Pediatric Drug Application; Jigsaw; Metaverse; Classical Education

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group 1 (Experimental): Intervention
  Interventions: Other: Jigsaw
- Intervention Group 2 (Experimental): Intervention
  Interventions: Other: Metaverse
- Control Group (Experimental): Control Group
  Interventions: Other: Classical Education

INTERVENTIONS:
Other: Jigsaw — In this learning method, students will be divided into main and expert groups. Then, an expert from each group will come and the student will be provided with expertise in the subject given to him/her by the instructor. After the student has specialized, he/she will return to his/her own group and will provide training to his/her friends on the subject he/she has specialized in under the supervision of the instructor of the course. During the student's specialization process on the subject given, the necessary literature support and controls will be provided by the instructor of the course.
  Arms: Intervention Group 1
Other: Metaverse — In this learning method, the topics determined on pediatric drug applications will be prepared weekly by the relevant instructor of the course and will be transferred to the metaverse and presented to the student in the form of weekly modules.
  Arms: Intervention Group 2
Other: Classical Education — In this learning method, the subjects determined by the instructor will be explained to the students in a laboratory environment by the instructor using a presentation (power point) method.
  Arms: Control Group

SUMMARY:
The aim of this study was to evaluate the effectiveness of jigsaw, metaverse and classical learning models in developing self-efficacy in medication administration of students taking pediatric nursing courses.

DETAILED DESCRIPTION:
Purpose of the Study The purpose of this study is to evaluate the effects of three different learning methods (classical, metaverse, jigsaw) used in pediatric drug application skills training on students' drug application self-efficacy levels in children.

Research Hypotheses H0: There is no difference between the drug application self-efficacy levels of students in groups.

H1: There is a difference between the drug application self-efficacy levels of students in groups.

Research Form This study is a pre-test post-test randomized quasi-experimental study. In addition, when the study is completed, a qualitative interview will be conducted with 10 volunteer students in each group regarding the positive and negative aspects of the classical, jigsaw and metaverse techniques.

Place and Time of the Study The study will be conducted with students taking the Child Health and Diseases Nursing Course of the Nursing Department of the Faculty of Health Sciences at Süleyman Demirel University between April and June 2023.

The Universe and Sample of the Study The universe of the study consists of 180 students taking the Nursing Department Child Health and Diseases Nursing Course. The 90 students determined as a result of the power analysis will be formed.

Power Analysis: The power analysis of the study was performed with the GPower 3.1.9.2. (Universitaet Kiel, Germany) program. Since the study design was prepared as three independent groups and two repeated measures, "F test" was selected as the test family and "ANOVA: Repeated measures, within-between interaction" was selected as the analysis. First of all, according to the main mass information given as N=180 with the single sample ratio test, the sample size was calculated as n=63 for the p=0.40 ratio value, 5% error and 95% power value. The effect size for the variance explained by the effect for repeated measures was calculated as d=0.252 for 1. The total sample size was calculated as n=66 for three independent groups and two repeated measurements under the conditions of 5% margin of error, 0.95 power value, and r=0.5 correlation between repeated measurements. However, considering the randomization and repeated study situation, it was decided to increase the sample slightly and complete it with 30 students for each group, totaling n=90.

Criteria for inclusion in the study:

* Being a first-time student taking the Child Health and Diseases Nursing Course
* Being a volunteer to participate in the study

Criteria for exclusion from the study:

* Being a Health Vocational High School graduate or being included in the program with DGS (vertical transfer exam)
* Not being a non-resident during the dates when the data of the study were collected
* Having received education or courses on drug applications in children in previous periods
* Being a student taking the course from below Randomization: Students who meet the criteria for inclusion in the study will be assigned to groups with the simple randomization method (classic, metaverse, jigsaw learning). Students who do not accept to participate in the research will receive the same topic from the relevant instructor in accordance with the routine of the course.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Child Health and Disease Nursing Course for the first time
* Volunteering to participate in the research

Exclusion Criteria:

* Not doing any treatment during the dates when the research data was collected
* Not taking any training or courses on drug applications in children in previous periods
* Not taking the course from the bottom

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pediatric medication administration self-efficacy scale score | 4 month
  The self-efficacy scale for medication administration in children for nursing students was developed by Bektaş et al. in 2021. The scale consists of 16 items and two sub-dimensions. The medication preparation sub-dimension for children (items for calculating and obtaining medication doses) is items 1, 2, 3, 4, 5, 6, 7, and 8; the medication administration sub-dimension (items for administering the obtained medication) is items 9, 10, 11, 12, 13, 14, 15, and 16. This scale is graded in a 5-point Likert-type scale and is listed as 1 = Definitely not sufficient, 2 = Somewhat sufficient, 3 = Partially sufficient, 4 = Sufficient, 5 = Definitely sufficient. The lowest score obtained from the scale is 16 and the highest score is 80. The scale has no cut-off point; as the score increases, the students' self-efficacy for pediatric medication administration increases. The scale has no reverse-scored items.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Nursing Department, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We can share all the details once our research is published.